CLINICAL TRIAL: NCT06633601
Title: A Prospective, Single-Centre, Single-Arm, Non-Randomized, Phase-I, MRI-Guided Ultrasound Stimulated Microbubbles Radiation Treatment for Patients with Chest-Wall and Locally Advanced Breast Cancer - a Pilot Study
Brief Title: MRI-Guided Ultrasound Stimulated Microbubbles Radiation Treatment for Patients with Chest-Wall and Locally Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Terry Fox Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5767
Record Dates: First submitted 2024-01-05; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Focused Ultrasound; Breast Cancer; Microbubbles
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Microbubbles

STUDY DESIGN:
Intervention Model Description: Experimental Arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): All biopsy confirmed breast cancer patients undergoing MRI-Ultrasound Stimulated Microbubble Radiation Treatment plus Radiation Therapy.
  Interventions: Device: MR-Guided Focused Ultrasound Technology; Drug: Definity Suspension for Injection

INTERVENTIONS:
Device: MR-Guided Focused Ultrasound Technology — MRI Guidance for use with High-intensity-focused ultrasound (HIFUS)
  Other Names: Arrayus System
Drug: Definity Suspension for Injection — Microbubble contrast agents for ultrasound
  Other Names: Microbubbles

SUMMARY:
The objective of this study is to demonstrate the feasibility of novel Magnetic Resonance Imaging (MRI)-guided ultrasound stimulated microbubble treatment to enhance radiation effects in humans receiving external beam radiotherapy delivered using a LINAC (linear accelerator) radiation therapy device.

DETAILED DESCRIPTION:
This is a prospective, single-centre, single-arm, non-randomized phase one (Phase I) clinical trial. In this study, locally advanced breast cancer (LABC) and breast/chest wall tumours not managed by surgery, patients will receive MRI-guided ultrasound-stimulated microbubble-treatment using an Arrayus MRI-FUS System combined with radiotherapy on a LINAC. Patients will lie on the MRI table with an in-built focused ultrasound platform where the tumour is kept in close contact with the transducer of the ultrasound. After exposure to the tumour with focused ultrasound, the patient will receive a standard of care LINAC-based radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* All biopsy-confirmed invasive ductal, invasive lobular and other rare histologic types of carcinoma.
* Patients with early stage Breast cancer, or LABC ; i.e., Stage IIA - IIIC cancers (T2 N0 M0 to Any T, N3, M0) or Stage IV (Any T, Any N, M1) per AJCC guidelines (8th Edition).
* Assessed as indicated, by a multidisciplinary team of treating medical, surgical and radiation oncologist and found suitable for radiation treatment.
* Patient referred for standard palliative radiotherapy or curative radiotherapy, which may include (but are not limited to) any of the following dose regimens: 1) 5-8 Gy in one fraction, 2) 20 Gy in 5 fractions, 3) 30 Gy in 5 fractions, 4) 35 Gy in 5 fractions, 5) 30 Gy in 10 fractions, 6) 40 Gy in 10 fractions, 5) 50 Gy in 20 fractions, 6) 60 Gy in 30 fractions and 7) 66 Gy in 33 fractions, or radiobiologically similar doses.
* Able to understand and give informed consent.
* Weight < 140 kg.
* Target lesion accessible for MRg-FUS+MB procedure.
* Able to communicate sensation during the procedure.
* Creatinine within normal institutional limits or creatinine clearance >60mL/min/ Novel MRI-Guided Ultrasound Stimulated Microbubble Radiation Treatment for Patients with Chest-Wall and Locally Advanced Breast Cancer. 1.73m2 for patients with creatinine levels above institutional upper limit of normal.

Exclusion Criteria:

* Pregnant or lactating women may not participate due to the embryotoxic effects of protocol treatment.
* Unable to have a contrast-enhanced MRI scan - standard of care criteria.
* Patients having received anthracycline or taxane based chemotherapy within the past 5 days.
* Patients with metallic or breast implants.
* Subjects with connective tissue disorder, musculoskeletal deformity.
* Target lesion causing deep ulceration, bleeding or discharge of the overlying skin.
* A fibrotic scar along the proposed FUS beam path.
* Severe cardiovascular, neurological, renal or hematological chronic disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥ 3.
* Any condition that in the investigator's opinion precludes participation.
* Unable to tolerate required stationary position during treatment.
* Allergy to Definity microbubbles.
* Cardiac disease or unstable hemodynamics including myocardial infarction within six months, unstable angina, congestive heart failure, cardiac shunts, cardiac arrhythmia and cardiac pacemaker.
* Contraindication to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation like cisapride, erythromycin, tricyclic antidepressants, Class IA and III antiarrhythmic agents and some antipsychotics like haloperidol, droperidol, quetiapine, thioridazine, ziprasidone.
* Known QT prolongation = (QTc > 450ms for men or >470ms for women) with cardiac impairment if ECG is requested as per SOC.
* History of bleeding disorder, coagulopathy.
* Severely impaired renal function with estimated glomerular filtration rate < 30ml/min/1.73m2 and/or on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety profile of MRI- guided ultrasound stimulated microbubble treatment and radiation in patients with inoperable breast/chest wall tumours or LABC. | 2 years
  The primary aim of this research is to evaluate the safety profile of MRI- guided ultrasound stimulated microbubble treatment and radiation in patients with inoperable breast/chest wall tumours or LABC.Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Tumour size response to MRg-FUS + MB and radiation, as measured radiologically or clinically within the treated therapeutic regions. | 2 years
  The secondary aim of this research is to evaluate tumour response to MRg-FUS + MB and radiation, as measured radiologically or clinically within the treated therapeutic regions. Outcomes will be measured using RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Czarnota, MD, PhD., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No